CLINICAL TRIAL: NCT03354520
Title: Optimizing Treatment Effects on OSA-related Clinical and Patient-centered Outcomes Among Blacks
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI departure from institution
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-01097
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tailored Videos (Active Comparator)
  Interventions: Behavioral: Tailored Videos
- Standard Videos (Active Comparator)
  Interventions: Behavioral: Standard Videos
- OSA Treatment (Active Comparator)
  Interventions: Behavioral: OSA Treatment

INTERVENTIONS:
Behavioral: Tailored Videos — web-based OSA messages (videos featuring role models and coaching advice using motivational enhancement) addressing OSA barriers within a health literacy framework--to decrease cognitive load and render messages understandable and actionable. OSA messages were tailored based on focus group data in the previous study (group tailoring).
  Arms: Tailored Videos
Behavioral: OSA Treatment — Web-based platform delivering messages promoting OSA self-efficacy. . All patients will view the introductory video, followed by the video cluster: Sleep, Health, and Well-Being; Sleep-Heart Health; Lifestyle Changes; and Sleep Hygiene.
  Arms: OSA Treatment
Behavioral: Standard Videos — Patients in the control arm will also receive an iPad, providing access to standard online OSA health information (e.g., National Sleep Foundation) in an equivalent dose as in the intervention arm using pre-selected automatic alerts to access the website
  Arms: Standard Videos

SUMMARY:
The study is to maximize efficacy of message delivery to achieve desired Obstructive sleep apnea (OSA) adherence goal. Newly diagnosed black patients (n=390, all genders) from participating sleep clinics will be randomly exposed to either the individually tailored or standard OSA messages. Investigators will look at an effective and scalable intervention to improve OSA-related outcomes: a) clinical CVD and brain health measures and b) patient-centered outcomes. Patient-centered and adherence data will be captured via REDCap, enabling real-time application of data-driven decision rules while implementing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported race/ethnicity as African American, African, Caribbean or black
* Accessible by phone
* No plans to move away within the year
* OSA diagnosis, consent, including permission to release medical data
* Physician-diagnosed medical conditions.

Exclusion Criteria:

* Progressive illnesses in which disability or death is expected within 1 year
* Impaired cognitive/ functional ability precluding participation
* Intention to move within the same year of enrollment
* Family member currently enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline OSA Self-Efficacy Scale Score to 6 Months Score | 2 Months and 6 Months
  The mean of the nonmissing item responses was calculated for each of the 3 subscales: Perceived Risk, Outcome Expectancies, and Treatment Self-Efficacy. Using this mean-weighted score prevents the distortion of the score from missing responses. Factor 1 (Risk Perception consisting of 8 questions); Factor 2 (Outcome Expectancy consisting of 9 items) and Factor 3 (Treatment Self Efficacy consisting of 9 items) are given a potential score of 1-4.

CONTACTS AND LOCATIONS:
Overall Officials: Girardin Jean-Louis, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Requests should be directed to Ferdinand.Zizi@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.